CLINICAL TRIAL: NCT00967369
Title: A Randomized Phase II Study of Bortezomib Plus ICE (BICE) Versus Standard ICE for Patients With Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Combination Chemotherapy With or Without Bortezomib in Treating Patients With Classical Hodgkin Lymphoma That Has Returned or Does Not Respond to Prior Treatment.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0604; NCI-2018-02154 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0604 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Recurrent Classic Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma
MeSH Terms: interventions — Bortezomib; Carboplatin; Etoposide; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (bortezomib, ifosfamide, carboplatin, etoposide) (Experimental): ARM A: Patients receive bortezomib IV over 5 seconds on days 1 and 4, ifosfamide IV continuously over 24 hours on day 1, carboplatin IV over 1 hour on day 1, and etoposide IV over 2 hours on days 1-3. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide
- Arm B (ifosfamide, carboplatin, etoposide) (Active Comparator): Patients receive ifosfamide, carboplatin and etoposide as in Arm A. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
  Arms: Arm A (bortezomib, ifosfamide, carboplatin, etoposide)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942

SUMMARY:
This phase II trial studies how well combination chemotherapy with or without bortezomib works in treating patients with classical Hodgkin lymphoma that has come back or does not respond to prior treatment. Drugs used in chemotherapy, such as ifosfamide, carboplatin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bortezomib is designed to block a protein that plays a role in cell function and growth. Bortezomib may cause cancer cells to die. It is not yet known if combination chemotherapy with or without bortezomib may work better in treating patients with classical Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate (ORR), partial remissions (PR), and complete remissions (CR) after 3 cycles of bortezomib plus ifosfamide, carboplatin, and etoposide (ICE) (BICE) versus ICE in patients with relapsed/refractory classical Hodgkin lymphoma (cHL).

II. To evaluate 2-year progression-free survival (PFS) in patients treated with 3 cycles of BICE versus ICE.

SECONDARY OBJECTIVES:

I. To compare positron emission tomography (PET) scan response after 3 cycles of BICE versus ICE chemotherapy.

II. To compare serum levels of tumor necrosis factor (TNF) proteins (a proliferation-inducing ligand [APRIL], B lymphocyte stimulator [BLyS], soluble [s]CD30, and CD40L) and CC thymus and activation-related cytokine (TARC) at baseline and after 3 cycles of BICE versus ICE chemotherapy.

III. To correlate baseline cytokine/chemokine levels with response to therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive bortezomib intravenously (IV) over 5 seconds on days 1 and 4, ifosfamide IV continuously over 24 hours on day 1, carboplatin IV over 1 hour on day 1, and etoposide IV over 2 hours on days 1-3. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive ifosfamide, carboplatin and etoposide as in Arm A. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory classical Hodgkin lymphoma.
* Patients must have received a front-line standard anthracycline-containing regimen, such as adriamycin-bleomycin-vinblastine-dacarbazine (ABVD), Stanford V, or bleomycin-etoposide-adriamycin-cyclophosphamide-oncovin-procarbazine-prednisone (BEACOPP).
* Bi-dimensionally measurable disease with at least 1 lesion >= 2.0 cm in a single dimension.
* Absolute neutrophil count (ANC) >= 1,500/microL.
* Platelet count >= 100,000/ microL.
* Hemoglobin >= 8 g/dL.
* Serum bilirubin < 2.0 mg/dL.
* Alkaline phosphatase < 2 x upper limits of normal (ULN).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 x ULN.
* Serum creatinine =< 1.5 mg/dL.
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2.
* Females of childbearing potential must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test and must agree to use 2 highly effective contraceptive methods (hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study and for 3 months after completion of protocol treatment. Females of non-childbearing potential are those who are postmenopausal for greater than 1 year or whom have had a bilateral tubal ligation or hysterectomy.
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 3 months after completion of protocol treatment.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Lymphocyte predominant Hodgkin lymphoma histology.
* More than one prior chemotherapy regimen.
* Prior autologous or allogeneic stem cell transplant.
* Presence of central nervous system (CNS) involvement with Hodgkin lymphoma.
* Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
* Active hepatitis B or C infection or history of cirrhosis.
* Grade 2 or greater peripheral neuropathy within 14 days of enrollment.
* Hypersensitivity to boron or mannitol.
* Prior bortezomib therapy.
* Another primary malignancy (other than squamous cell and basal cell carcinoma of the skin, in situ carcinoma of the cervix, or squamous intraepithelial lesion on PAP smear, or treated prostate cancer with a stable prostate specific antigen [PSA]) for which the patient has not been disease-free for at least 3 years.
* Patients with congestive heart failure, Class III or IV, by New York Heart Association (NYHA) criteria.
* Patients with a myocardial infarction 6 months prior to enrollment, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiogram (ECG) evidence of acute ischemia or active conduction system abnormalities.
* Patient with other medical or psychiatric illness that is likely to interfere with participation in this clinical study.
* Female subject that is pregnant or breast-feeding.
* Patient that has received other investigational drugs within 14 days of enrollment.
* Patients using concurrent therapy with corticosteroids at greater than or equal to 20 mg/day of prednisone equivalent.
* Patients with active systemic bacterial, viral, or fungal infections that have required IV antimicrobials within 4 weeks prior to protocol treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08-24 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Fanale, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 2009 to August 2011 at MD Anderson Cancer Center.
Groups:
- BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide); ICE (Ifosfamide, Carboplatin, Etoposide): Relapsed/refractory classical Hodgkin lymphoma who have received a front-line standard anthracycline-containing regimen, such as ABVD, Stanford V, or BEACOPP.
Period: Overall Study
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide)
Started | 10 | 10
Relapsed | 4 | 7
Refractory | 6 | 3
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
  Mexico | 1 | 0 | 1
A Randomized Phase II Study of Bortezomib Plus ICE (BICE) Versus Standard ICE for Patients with Rela [Count of Participants; unit: Participants]
  Mobilization regimens:Ifosfamide +etoposide | 7 | 8 | 15
  Mobilization regimen:Gemcitabine,Navelbine,Doxorub | 2 | 1 | 3
  Mobilization regimen:Cyclophosphamide | 1 | 0 | 1
  SD by CT imaging, but given PET negativity, receiv | 0 | 1 | 1
  Conditioning regimen Gemcitabine/Busulfan/melphala | 9 | 9 | 18
  Conditioning regimen BEAM followed with ASCT | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response After 3 Cycles of Botezomib Plus ICE (BICE) Versus Ifosfamide, Carboplatin, Etoposide (ICE) in Patients With Relapsed/Refractory Classical Hodgkin Lymphoma
Description: Response rates for Bortezomib, Ifosfamide, Carboplatin, Etoposide (BICE) and Ifosfamide, Carboplatin, Etoposide (ICE) treatment groups were assessed by the 1999 International Working Group (IWG)(CT alone) (Cheson et al., 1999) and compared to 2007 IWG (CT plus PET) (Cheson et al., 2007) criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From baseline to 3 cycles of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide)
Number analyzed (Participants) | 10 | 10
Participants
  Overall Response | 7 | 6
  Complete Response (CR) | 3 | 1
  Partial Response (PR) | 4 | 5
  Progressive Disease (PD) | 0 | 0
  Stable Disease (SD) | 1 | 3

2. Primary Outcome: Progression Free Survival (PFS) Rate at 12 Months
Description: Progression free survival time is defined as the time interval from treatment start to progression or death due to any cause whichever happens first. Participants will be censored at the last follow-up date, if an event(progression/death) is not observed during the follow-up.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Measure: Number; unit: percentage of participants
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide)
Number analyzed (Participants) | 10 | 10
percentage of participants | 50 | 70

3. Primary Outcome: Overall Survival (OS) Rate at 24 Months
Description: Overall Survival is time from date of treatment start until date of death due to any cause or last Follow-up within 24 months.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide)
Number analyzed (Participants) | 10 | 10
percentage of participants | 70 | 89

4. Secondary Outcome: PET Scan Response After 3 Cycles of BICE Versus ICE Chemotherapy.
Description: Response rates for BICE and ICE treatment groups will be assessed by 1999 IWG (CT alone) (Cheson et al., 1999) and compared to 2007 IWG (CT plus PET) (Cheson et al., 2007) criteria.
Time Frame: Baseline up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide)
Number analyzed (Participants) | 10 | 10
Participants
  PET negativity : Complete Response (CR) | 3 | 6
  PET negativity : Partial Response (PR) | 0 | 4
  PET negativity : Stable Disease (SD) | 0 | 1
  PET positivity : Partial Response (PR) | 4 | 2
  PET positivity : Stable Disease (SD) | 1 | 2
  PET positivity : Progressive Disease (PD) | 2 | 0

5. Secondary Outcome: Serum Levels of Tumor Necrosis Factor (TNF) Proteins (APRIL, BLyS, sCD30, and CD40L) and CC Thymus and Activation-related Cytokine (TARC) at Baseline and After 3 Cycles of BICE Versus ICE Chemotherapy
Time Frame: November 2009 and December 2010
Population: Incomplete report as study was stopped early due to futility
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Baseline Cytokine/Chemokine Levels With Response to Therapy.
Time Frame: 106 weeks/13 months/426 days
Population: Incomplete report as study was stopped early due to futility. Participant with relapsed/refractory HL prior to autologous transplant
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) | ICE (Ifosfamide, Carboplatin, Etoposide)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) (N=10) | ICE (Ifosfamide, Carboplatin, Etoposide) (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BICE (Bortezomib, Ifosfamide, Carboplatin, Etoposide) (N=10) | ICE (Ifosfamide, Carboplatin, Etoposide) (N=10)
Neutrophil count decreased (Investigations) | 7 | 5
Platelet count decreased (Investigations) | 7 | 5
Transaminitis (Investigations) | 8 | 5
Hyperbilirubinemia (Investigations) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-06-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT00967369/Prot_SAP_000.pdf